CLINICAL TRIAL: NCT04707300
Title: A Phase I/II Study Evaluating the Safety and the Efficacy of Human T Lymphoid Progenitor (HTLP) Injection to Accelerate Immune Reconstitution After Umbilical Cord Blood (UCB) Transplantation in Adult Patients With Hematologic Malignancies
Brief Title: Study Evaluating the Safety and the Efficacy of Human T Lymphoid Progenitor (HTLP) Injection to Accelerate Immune Reconstitution After Umbilical Cord Blood (UCB) Transplantation in Adult Patients With Hematologic Malignancies (HTLP-ONCO)
Acronym: HTLP-ONCO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP191116; 2019-004883-23 (EudraCT Number)
Record Dates: First submitted 2020-11-30; First posted 2021-01-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Malignancy
Keywords: acute myeloid leukemia; minimal residual disease; hematologic malignancies; human T Lymphoid Progenitor; umbilical cord blood transplantation
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human T Lymphoid Progenitor (HTLP) injection (Experimental): HTLP cellular product obtained after 7 days of culture of immune-selected CB
  Interventions: Drug: Human T Lymphoid Progenitor (HTLP) injection

INTERVENTIONS:
Drug: Human T Lymphoid Progenitor (HTLP) injection — The HTLP cell suspension will be injected intravenously at the time of UCB HSCT on D0

SUMMARY:
This is an open-labelled and non-controlled Phase I/II clinical trial, evaluating the safety and the efficacy of Human T Lymphoid Progenitor (HTLP) injection to accelerate immune reconstitution after umbilical cord blood (UCB) transplantation in adult patients with hematologic malignancies. The dose limiting toxicity of HTLP injection will be evaluated using a model-based design.

DETAILED DESCRIPTION:
Allogeneic bone marrow transplantation (AlloSCT) is the treatment of choice for high- risk acute myeloid leukemias in complete first remission after induction therapy and other high-risk hematological malignancies. Umbilical cord blood grafts are frequently used for patients lacking an HLA- matched family donor (Matched-sibling donor, MSD) as well as in the absence of an appropriate unrelated donor (10/10 MUD). As any HSCT, UCB transplantations are associated with the risk of acute and chronic GVHD, post- transplant immunodeficiency with increased risk of infections as well as relapse. Especially the risk of infection and therefore non- relapse mortality (NRM) or transplant- related mortality (TRM) is significantly higher in UCB transplantations as compared to MSD or 10/10 MUD transplantations. All of these risks have been linked to a significant delay in immune reconstitution including various immune cell populations like CD4 and CD8 T cells, Treg, NK, iNKT, pDC and others.

The investigators therefore make the hypothesis that if T-cell-mediated immunity was rapidly generated after a partially HLA-compatible UCB transplantation will reduce the risk of infection and to prevent relapse without increasing the risk of GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old and <66 years old) at the time of inclusion and eligible for an allogeneic stem cells transplantation and fit to receive the specified conditioning regimen
* Patients with hematologic malignancies
* Absence of a matched - related sibling donor (MSD) or a matched unrelated donor (MUD) 10/10
* Presence of two UCB units with the following criteria*: HLA- matched 4/8, 5/8, 6/8, 7/8 or 8/8 for HLA- A, -B, -C and DRB1 loci

AND

• Presence of at least one UCB unit with the following criteria*: ≥ 3 x 10e7 TNC/kg or ≥ 1.5 10e5 CD34+/kg pre- freezing

* For the UCB taken into HTLP culture, the CD34+ content does not need to meet the above cellularity criteria, as expansion during HTLP culture has been proven to ensure the appropriate number of CD7+ needed for each dose.

The non- cultured UCB will be chosen to have a higher CD34+ cell content in order to enable long- term hematopoietic engraftment

* Absence of Donor Specific Antibodies (DSA) with a MFI > 5000
* Patient affiliated to social security
* Written, informed consent of the patient

Exclusion Criteria:

* Any of the standard contraindications to allogeneic transplant
* Left ventricular ejection fraction <50%
* Abnormal biochemistry results (ALT/AST>10xULN, total bilirubin>2.5xULN, creatinin clearance <60ml/min)
* Inability to understand and provide informed consent
* Concomitant infectious disease: HTLV-I, HIV-I or HIV-II
* Pregnancy or breastfeeding for women of childbearing potential
* Patients with progressive hematologic malignancies
* Previous participation within one month before inclusion in another protocol in which drugs may influence immune reconstitution of bone marrow transplantation

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of grade III-IV graft-versus-host disease (GvHD) | Within 100 Days following HSCT
  according to Glucksberg grading system, to define toxicity
CD4 + T cells analysis | Within 100 days following HSCT
  Efficacy defined by the presence of >50/μl CD4+ CD3+ TCRαβ+ T cells at 2 consecutive measures < within 4 months post HSCT.

SECONDARY OUTCOMES:
Time to hematologic engraftment | Up to 24 months post-transplantation
  ANC > 0.5G/L and platelets > 20G/L on 3 consecutive days
Last transfusion of platelets and red blood cell | During the follow-up
Absolute numbers of neutrophils | Month 1, 2, 3, 6 and 12 post -transplantation
Time course of T cell immune reconstitution | Month 1, 2, 3, 6 and 12 post -transplantation
  by immunophenotyping (flow cytometry analysis) - with a focus on time needed to exceed a count of 100 naive CD4+ and >100 total CD8+ cells per μL
Immune phenotype (flow-cytometry analysis) of the different TCRαβ+ cell subpopulations | Month 1, 2, 3, 6 and 12 post -transplantation
  TCD4 naive/memory population (CD31+CD45RA+/CD4+, CD45RO/CD4+; CD31+CD4+); TCD8 naive/memory population (CD45RA+CCR7+/CD8+, CD45RA-CCR7+/ CD8+, CD45RA- CCR7+/ CD8+, CD45RA-CCR7-/CD8+) , CD8 effector memory RA+ (TEMRA) (CD45RA+CCR7- /CD8+ ); Regulatory T cells (CD4+CD25+CD127lowCD25+).
  • Analysis of CD3, CD4, CD8 numbers will be performed if total lymphocytes ≥ 500/μL and analysis of T cell subpopulations if CD3+ cells ≥ 1000/μL
B-cell reconstitution | Month 1, 2, 3, 6 and 12 post -transplantation
  (B CD19 naive/memory population (CD27-IgD+/CD19+, CD27+IgD+/CD19+, CD27+IgD-/CD19 and Ig levels) at 1, 2, 3, 6 and 12 months post HSCT with focus on time needed for cessation of intravenously IgG replacement therapy
Reconstitution of the NK cell | Month 1, 2, 3, 6 and 12 post -transplantation
  compartment (CD16+CD56+)
Assessment of engraftment of each UCB unit over time by hematological monitoring and chimerism analysis | at 1, 2, 3, 6 and 12 months following HSCT.
  at 1, 2, 3, 6 and 12 months following HSCT and between M1 and M2 post-transplantation if necessary according to the result of the chimerism at M1 on neutrophils, T, B, NK, pDC and macrophages.
  • The chimerism is studied on whole blood and on mononuclear cells (i.e. cells reconditioning after Ficoll) until the total number of lymphocyte is ≥ 100/μL.
  When lymphocyte count is ≥ 100/μL, the chimerism will be analysed on immunoselected cell populations (CD15+/CD3+/NK, CD19+)
Graft failure/rejection rate | at 3 months following HSCT
  detected by hematological monitoring of each UCB unit
Cumulative incidence of infections | at 3, 6 and 12 months post- transplantation
Cumulative incidence of acute and chronic episodes of GVHD and their grade according to Glucksberg GvHD staging. | at 3, 6, 12 and 24 months post-transplantation
Relapse rate | 2 years
Overall survival | 2 years
Disease-free survival | 2 years
Progression-free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HERMINE, PhD & MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Elisa MAGRIN, MD, Study Director — Département de Biothérapie : Hôpital Necker Enfants malades
Locations (5):
- France (5):
  - Hôpital Saint Louis, Paris
  - Service d'Hématologie et thérapie cellulaire / CHU of Bordeaux, Pessac
  - IUCT Oncopole Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif
  - Hematology department / Necker Children's Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No